CLINICAL TRIAL: NCT04727086
Title: Role of BP1.3656 on Alcohol Responses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 072/2017
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder
Keywords: Ethanol; Alcohol; Self administration; BP1.3656B; Alcohol Use Disorder; Alcoholism; Alcohol Drinking; Drinking Behavior; Alcohol-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Drinking Behavior; Alcohol-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This will be a within-subjects, counterbalanced, crossover trial with a washout period. Participants will receive either placebo or the interventional drug BP1.3656 during the initial 14-day phase of the study and receive the other intervention during the second 14-day phase of the study. The washout period will last a minimum of 14 days.
  Participants will come in to the laboratory on two separate days near the end of each intervention phase to complete alcohol self-administration sessions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication (BP1.3656) (Experimental): Participants will receive BP1.3656 in tablet form once daily at a dose of 30 µg/day for the first 4 days, followed by 60 µg/day for the remaining 10 days. If the highest dose is not tolerated, it will be lowered to 30 µg.
  Interventions: Drug: BP1.3656
- Placebo pills (Placebo Comparator): Participants will receive matching placebo pills for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP1.3656 — BP1.3656 will be administered in tablet form once daily at a dose of 30 µg/day for the first 4 days of the intervention phase, followed by a dose increase to 60 µg/day for the remaining 10 days. If the highest dose is not tolerated, it will be lowered to 30 µg.
  Arms: Medication (BP1.3656)
Drug: Placebo — Administered once daily in tablet form.
  Arms: Placebo pills

SUMMARY:
The current study will determine whether a novel pharmacotherapy, BP1. 3656, affects laboratory alcohol self-administration in participants with alcohol use disorder (AUD).

DETAILED DESCRIPTION:
The current study employs BP1.3656, a novel investigational compound with a track record for safety and tolerability in phase I clinical trials. When administered to mice, BP1.3656 was associated with increased metabolism of histamine and elevated brain dopamine and acetylcholine, suggestive of utility in psychiatric disorders including Alcohol Use Disorder (AUD).

This study is a Phase II laboratory-based trial of BP1 .3656 for AUD. 40 non-treatment seeking participants with AUD will be recruited. Participants will be randomly assigned to intervention with BP1 .3656 or placebo in a within-subject, crossover design. During each intervention period, outcome measures relating to alcohol motivation and self-administration will be assessed in the laboratory. It is hypothesized that relative to placebo, alcohol self-administration will be decreased by BP1 .3656.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling Diagnostic and Statistical Manual (DSM)-5 criteria for AUD with endorsement of 4-8 symptoms
* Average weekly consumption ≥ 14 standard drinks for women and ≥ 21 standard drinks for men over the past 3 months
* Willingness to take study medication and participate in laboratory sessions requiring alcohol administration
* Able to give written informed consent
* Certified as healthy by a comprehensive clinical assessment. Alanine transaminase (ALT) and aspartate aminotransferase (AST) levels should not be more than 1.2 times normal

Exclusion Criteria:

* Seeking treatment for alcohol use (or current efforts to cut down or seek treatment)
* A Clinical Institute Withdrawal Assessment (CIWA) score of 8+ upon initial assessment
* Current medical conditions or medications that contraindicate receiving the study drug (based on the study physician's assessment)
* Meeting criteria for a current substance use disorder aside from alcohol or nicotine
* Recent recreational drug use (assessed via urine toxicology screen)
* History of gross psychiatric or neurological impairment (e.g., schizophrenia, bipolar disorder, neurological disorders)
* Reported difficulty with intravenous procedures
* Self-report of significant alcohol-induced flushing after 1-2 drinks (a proxy for aldehyde dehydrogenase deficiency)
* Currently nursing or pregnant (females)
* Serious unstable medical condition
* Current use of medication that could increase the risk of BP1.3656B administration
* Having any clinical condition, drug sensitivity, or prior therapy which, in the investigator's opinion, makes the participant unsuitable for the study
* Any history of seizures

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Peak breath alcohol concentration (mg%) during free-access alcohol self-administration while taking study medication (BP1.3656). | Measured during one self-administration session in the 2nd week of the 14-day study medication phase.
  Breath alcohol concentration (BrAC) test reading will be assessed
Peak breath alcohol concentration (mg%) during free-access alcohol self-administration while taking placebo. | Measured during one self-administration session in the 2nd week of the 14-day placebo phase.
  Breath alcohol concentration (BrAC) test reading will be assessed
Motivation for alcohol completed during a progressive ratio alcohol self-administration session while taking study medication (BP1.3656). | Measured during one progressive-ratio self-administration session in the 2nd week of the 14-day medication phase
  Measured by number of button presses/work sets
Motivation for alcohol completed during a progressive ratio alcohol self-administration session while taking placebo. | Measured during one progressive-ratio self-administration session in the 2nd week of the 14-day placebo-phase.
  Measured by number of button presses/work sets

SECONDARY OUTCOMES:
Subjective effects of alcohol during free-access and progressive ratio self-administration sessions while taking study medication (BP1.3656), as measured by the Biphasic Alcohol Effects Scale (0-10 scoring) | Measured during each of two alcohol self-administration sessions (free-access, progressive ratio) completed in the 2nd week of the 14-day medication phase.
  Two subscales (stimulant and sedative) with a 0-10 scoring where higher scores for stimulant subscale indicate increased stimulated effects from alcohol, while higher scores for sedative subscale indicate more sedated effects from alcohol.
Subjective effects of alcohol (maximum reported stimulation and sedation from alcohol) during free-access and progressive ratio self-administration sessions while taking placebo, as measured by the Biphasic Alcohol Effects Scale (0-10 scoring) | Measured during each of two alcohol self-administration sessions (free-access, progressive ratio) completed in the 2nd week of the 14-day placebo phase.
  Two subscales (stimulant and sedative) with a 0-10 scoring where higher scores for stimulant subscale indicate increased stimulation, while higher scores for sedative subscale indicate more sedated effects from alcohol.
Self-reported craving after a priming dose of alcohol during free-access and progressive ratio self-administration sessions while taking BP1.3656, as measured by the Alcohol Urge Questionnaire (1-7 scoring) | Measured during each of 2 alcohol self-administration sessions (free-access, progressive ratio) completed in 2nd week of medication phase.
  8 statements with score options ranging from Score of 1 = Strongly disagree to Score of 7 = Strongly Agree. Higher scores reflect greater craving.
Self-reported craving after a priming dose of alcohol during free-access and progressive ratio self-administration sessions while taking placebo, as measured by the Alcohol Urge Questionnaire (1-7 scoring) | Measured during each of 2 alcohol self-administration sessions (free-access, progressive ratio) completed in 2nd week of placebo phase.
  8 statements with score options ranging from Score of 1 = Strongly disagree to Score of 7 = Strongly Agree. Higher scores reflect greater craving.
Safety and tolerability of BP1.3656 | During the free-access and progressive ratio sessions in the 2nd week of the 14-day study medication phase
  Side effects of BP1.3656 will be assessed with the Systematic Assessment for Treatment Emergent Effects questionnaire (not reporting score on a scale) and the Pittsburgh Sleep Quality Index (19 items with 0-3 scoring, where higher scores indicate worse sleep quality).
Safety and tolerability of BP1.3656 | During the free-access and progressive ratio sessions in the 2nd week of the 14-day study placebo phase
  Side effects of BP1.3656 will be assessed with the Systematic Assessment for Treatment Emergent Effects questionnaire (not reporting score on a scale) and the Pittsburgh Sleep Quality Index (19 items with 0-3 scoring, where higher scores indicate worse sleep quality).
Weekly alcohol consumption during treatment with BP1 .3656 | Measured during the 2nd week of the 14-day study medication phase
  Drinks per week, as measured by the Timeline Follow-Back method
Weekly alcohol consumption during treatment with placebo | Measured during the 2nd week of the 14-day placebo phase
  Drinks per week, as measured by the Timeline Follow-Back method

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No